CLINICAL TRIAL: NCT00368849
Title: Atomoxetine for Attention Deficits in Adults With Mild HD: A Randomized, Placebo-Controlled Crossover Study
Brief Title: Atomoxetine and Huntington's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Beglinger, Leigh J, Associate Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200508775
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2012-11-27 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Huntington Disease; Chorea
Keywords: Huntington Disease; Chorea; Attention; ADHD; ADD; Strattera; Atomoxetine
MeSH Terms: conditions — Huntington Disease; Chorea; Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 40 milligram twice a day atomoxetine (Experimental): Participants received 40 milligram twice a day atomoxetine for 4 weeks.
  Interventions: Drug: atomoxetine
- Twice a day matching placebo (Placebo Comparator): Participants received twice a day matching placebo for 4 weeks.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: atomoxetine — This study utilizes a crossover design. Accordingly, half of the participants receive 40 milligram twice a day atomoxetine at arm one while the remaining half receive this intervention at arm two.
  Other Names: Strattera
  Arms: 40 milligram twice a day atomoxetine
Drug: Matching Placebo — This study utilizes a crossover design. Accordingly, half of the participants receive twice a day matching placebo at arm one while the remaining half receive this intervention at arm two.
  Other Names: Sugar pill
  Arms: Twice a day matching placebo

SUMMARY:
The purpose of this research study is to evaluate the effect of atomoxetine (also known as Strattera) compared to placebo (inactive substance) on daily activities such as attention and focus, thinking ability and muscle movements in subjects with early Huntington Disease (HD) and attention deficit disorder (ADD).

DETAILED DESCRIPTION:
No medications have been investigated to improve attention and executive functions in patients with Huntington's disease, despite the evidence that these cognitive domains can be abnormal even before motor symptom onset. Because cognitive symptoms are highly associated with functional disability, treatments aimed at improving cognitive functions would be of significant benefit to patients in the early stages of the disease. Atomoxetine is the ideal choice for such a trial. It has proven efficacy in adults with attention deficit hyperactivity disorder (ADHD) and it selectively targets norepinephrine and dopamine in the prefrontal cortex rather than in subcortical areas. This selectivity is an advantage for patients with HD, because motor side effects are less likely to be facilitated than with a psychostimulant. The present study is a feasibility study in which we propose to administer either 80 milligram (mg) atomoxetine for 4 weeks or placebo to 20 patients with early HD who also complain of mild cognitive symptoms. The groups will then crossover to the other condition (atomoxetine or placebo). Participants will be assessed on measures of ADHD symptoms and a sensitive battery of neuropsychological tests. Based on the shared neural circuitry in ADHD and HD, and the demonstrated effectiveness of atomoxetine on attention in adults with ADHD, improved performance on cognitive tests of attention and executive functions and on subjects' report of ADHD symptoms are expected in the atomoxetine treatment phase. No changes in motor status are predicted during the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Huntington's disease (HD) diagnosis
* Age 18 to 65
* Must have mild HD
* Must have complaints of poor attention

Exclusion Criteria:

* Childhood history of attention deficit hyperactivity disorder (ADHD) symptoms
* Diagnosis of schizophrenia, bipolar affective disorder, dementia, delirium or severe anxiety
* Current use of a monoamine oxidase inhibitor (MAOI) medication
* Pregnancy
* Uncontrolled hypertension
* Tachycardia
* Cardiovascular or cerebrovascular disease
* History of a loss of consciousness for greater than (or equal to) 5 minutes
* Having any neurological disorder or insult other than Huntington disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh J Beglinger, Ph.D., Principal Investigator — University of Iowa
Locations (1):
- The University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Background] A novel gene containing a trinucleotide repeat that is expanded and unstable on Huntington's disease chromosomes. The Huntington's Disease Collaborative Research Group. Cell. 1993 Mar 26;72(6):971-83. doi: 10.1016/0092-8674(93)90585-e. PMID 8458085
- [Background] Campodonico JR, Aylward E, Codori AM, Young C, Krafft L, Magdalinski M, Ranen N, Slavney PR, Brandt J. When does Huntington's disease begin? J Int Neuropsychol Soc. 1998 Sep;4(5):467-73. doi: 10.1017/s1355617798455061. PMID 9745236
- [Background] Lawrence AD, Hodges JR, Rosser AE, Kershaw A, ffrench-Constant C, Rubinsztein DC, Robbins TW, Sahakian BJ. Evidence for specific cognitive deficits in preclinical Huntington's disease. Brain. 1998 Jul;121 ( Pt 7):1329-41. doi: 10.1093/brain/121.7.1329. PMID 9679784
- [Background] Paulsen JS, Zhao H, Stout JC, Brinkman RR, Guttman M, Ross CA, Como P, Manning C, Hayden MR, Shoulson I; Huntington Study Group. Clinical markers of early disease in persons near onset of Huntington's disease. Neurology. 2001 Aug 28;57(4):658-62. doi: 10.1212/wnl.57.4.658. PMID 11524475
- [Background] Marder K, Zhao H, Myers RH, Cudkowicz M, Kayson E, Kieburtz K, Orme C, Paulsen J, Penney JB Jr, Siemers E, Shoulson I. Rate of functional decline in Huntington's disease. Huntington Study Group. Neurology. 2000 Jan 25;54(2):452-8. doi: 10.1212/wnl.54.2.452. PMID 10668713
- [Background] Gomez-Tortosa E, MacDonald ME, Friend JC, Taylor SA, Weiler LJ, Cupples LA, Srinidhi J, Gusella JF, Bird ED, Vonsattel JP, Myers RH. Quantitative neuropathological changes in presymptomatic Huntington's disease. Ann Neurol. 2001 Jan;49(1):29-34. PMID 11198293
- [Background] Beglinger, L. et al. The association between speed of processing and cerebral white matter volume in patients with mild Huntington's disease [abstract]. Poster session accepted at the Annual Meeting of the Cognitive Neuroscience Society, April, 2004
- [Background] Halliday GM, McRitchie DA, Macdonald V, Double KL, Trent RJ, McCusker E. Regional specificity of brain atrophy in Huntington's disease. Exp Neurol. 1998 Dec;154(2):663-72. doi: 10.1006/exnr.1998.6919. PMID 9878201
- [Background] Nopoulos, P. et al., (under review). Structural Brain Abnormalities in pre-symptomatic Huntington's disease.
- [Background] Aylward EH, Anderson NB, Bylsma FW, Wagster MV, Barta PE, Sherr M, Feeney J, Davis A, Rosenblatt A, Pearlson GD, Ross CA. Frontal lobe volume in patients with Huntington's disease. Neurology. 1998 Jan;50(1):252-8. doi: 10.1212/wnl.50.1.252. PMID 9443488
- [Background] Casey BJ, Castellanos FX, Giedd JN, Marsh WL, Hamburger SD, Schubert AB, Vauss YC, Vaituzis AC, Dickstein DP, Sarfatti SE, Rapoport JL. Implication of right frontostriatal circuitry in response inhibition and attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 1997 Mar;36(3):374-83. doi: 10.1097/00004583-199703000-00016. PMID 9055518
- [Background] Hale TS, Hariri AR, McCracken JT. Attention-deficit/hyperactivity disorder: perspectives from neuroimaging. Ment Retard Dev Disabil Res Rev. 2000;6(3):214-9. doi: 10.1002/1098-2779(2000)6:33.0.CO;2-M. PMID 10982499
- [Background] Heilman KM, Voeller KK, Nadeau SE. A possible pathophysiologic substrate of attention deficit hyperactivity disorder. J Child Neurol. 1991;6 Suppl:S76-81. doi: 10.1177/0883073891006001s09. PMID 2002218
- [Background] Spencer T, Biederman J, Wilens T, Prince J, Hatch M, Jones J, Harding M, Faraone SV, Seidman L. Effectiveness and tolerability of tomoxetine in adults with attention deficit hyperactivity disorder. Am J Psychiatry. 1998 May;155(5):693-5. doi: 10.1176/ajp.155.5.693. PMID 9585725
- [Background] Michelson D, Adler L, Spencer T, Reimherr FW, West SA, Allen AJ, Kelsey D, Wernicke J, Dietrich A, Milton D. Atomoxetine in adults with ADHD: two randomized, placebo-controlled studies. Biol Psychiatry. 2003 Jan 15;53(2):112-20. doi: 10.1016/s0006-3223(02)01671-2. PMID 12547466
- [Background] Conners, CK et al. Conners' Adult ADHD Rating Scales (CAARS). 1999. North Tonawanda, NY: Multi-Health Systems.
- See also: University of Iowa Huntington's Disease Center of Excellence — http://www.uihealthcare.com/depts/huntingtonsdisease/index.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (number = 20) were recruited using advertisements and through the University of Iowa Huntington Disease (HD) Registry at a rate of 1.40 individuals per month from September 2006 through November 2007 (i.e., 14.3 months).
Pre-assignment Details: Participants were screened before baseline for the presence of attentional problems through interview, medical status (including safety laboratories and electrocardiogram), and history for inclusion/exclusion criteria.
Groups:
- Atomoxetine (4 Weeks) Then Placebo (4 Weeks): Participants received 40 milligram twice a day atomoxetine for four weeks. After a two week wash out, they then received twice a day matching placebo for four weeks.
- Placebo (4 Weeks) Then Atomoxetine (4 Weeks): Participants received twice a day matching placebo for four weeks. After a two week washout, they then received 40 milligram twice a day atomoxetine for four weeks.
Period: Overall Study
Arm/Group | Atomoxetine (4 Weeks) Then Placebo (4 Weeks) | Placebo (4 Weeks) Then Atomoxetine (4 Weeks)
Started | 10 | 10
Completed | 10 | 8
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Age, sex, and region of enrollment were available for all 20 participants.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46.20 (10.288)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Conners' Adult Attention Rating Scale (CAARS)
Description: The Conners' Adult Attention Rating Scale (CAARS) is one of the most frequently used self-rating measures for adult Attention Deficit Hyperactivity Disorder (ADHD) and was given as a self-report measure of attention. It has 66 items with each item ranging from 0 to 3 points. Higher total scores represent greater impairment. The outcome reported was change in score from baseline for each treatment arm.
Time Frame: There are two time points for this measure: baseline and after 4 weeks of treatment
Population: Analysis was based on number of completers
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Atomoxetine: Individuals in this arm received 40 milligram twice a day atomoxetine
- Placebo: Individuals in this arm received twice a day matching placebo.
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 18 | 20
units on a scale | -2.88 (1.1) | -2.24 (1.1)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; The primary measures were analyzed as pretreatment and posttreatment difference scores using a series of analyses of covariance controlling for age. The results were screened for model violations (e.g., outliers). Preliminary analyses assured no treatment order effects by examining block by treatment interactions; Test type: Superiority or Other; p = 0.63, ANCOVA; Mean Difference (Final Values) = -0.65

2. Primary Outcome: Attention Composite Score
Description: The attention composite comprises performance on Wechsler Adult Intelligence Scale III Symbol-Digit and Letter Number Sequencing Subtests, Trail Making Test Part A, computerized simple-choice reaction time, and computerized working memory (i.e., 2-Back). The composite score is the average combined z score for each test. Higher, positive values indicate better than average performance and negative and lower values indicate worse than average. The outcome reported was change in score from baseline for each treatment arm.
Time Frame: There are two time points for this measure: baseline and after 4 weeks of treatment
Population: Analysis was based on number of completers.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 18 | 20
Units on a scale | -0.13 (0.07) | 0.02 (0.06)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.09, ANCOVA; Mean Difference (Final Values) = -0.15

3. Primary Outcome: Executive Composite Score
Description: The executive composite comprises performance on Trail Making Test Part B, Stroop Color and Word Test, and the Controlled Oral Word Association Test (i.e., Verbal Fluency). The composite score is the average combined z score for each test. Positive values indicate better than average performance and negative values worse than average. The outcome reported was change in score from baseline for each treatment arm.
Time Frame: There are two time points for this measure: baseline and after 4 weeks of treatment
Population: Analysis was based on number of completers.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 18 | 20
units on a scale | -1.68 (1.4) | -2.94 (1.4)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.46, ANCOVA; Mean Difference (Final Values) = 1.26

4. Secondary Outcome: Symptom Checklist-90-Revised (SCL-90-R)
Description: Psychiatric symptoms were evaluated with the Symptom Checklist-90-Revised, a self report measure of psychiatric symptoms. The measure produces raw scores and normed scores (T scores Mean = 50), with higher values representing greater impairment. The outcome reported was change in score from baseline for each treatment arm.
Time Frame: There are two time points for this measure: baseline and after 4 weeks of treatment
Population: Analysis was based on number of completers.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 18 | 20
units on a scale | -4.20 (1.9) | -4.64 (1.8)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; The secondary measures were analyzed as pretreatment and posttreatment difference scores using a series of analyses of covariance controlling for age. The results were screened for model violations (e.g., outliers). Preliminary analyses assured no treatment order effects by examining block by treatment interactions; Test type: Superiority or Other; p = 0.84, ANCOVA; Mean Difference (Final Values) = 0.44

5. Secondary Outcome: Unified Huntington Disease Rating Scale (UHDRS) Total Motor Score
Description: Although changes in motor symptoms were not hypothesized, the Unified Huntington Disease Rating Scale motor examination was administered at every visit. An experienced motor rater completes a motor examination and rates the participant on several motor tasks. Total score ranges from 0 - 124, with higher scores indicating a worse outcome. The outcome reported was change in score from baseline for each treatment arm.
Time Frame: There are two time points for this measure: baseline and after 4 weeks of treatment
Population: Analysis was based on number of completers.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 18 | 20
units on a scale | 0.42 (1.8) | -0.35 (1.7)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.76, ANCOVA; Mean Difference (Final Values) = 0.77

ADVERSE EVENTS:
Time Frame: Adverse events were reported from September 2006 through November 2007 (14.3 months)
Groups:
- Matching Placebo: Individuals in this arm received twice a day matching placebo.
Arm/Group | Atomoxetine | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 3/20
Other Adverse Events (participants affected / at risk) | 10/18 | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=20) | Matching Placebo (N=20)
Inpatient Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1)
An Important Medical Event (Renal and urinary disorders) | 0 (0) | 1 (1) — Elevated Creatinine Level
An Important Medical Event (Psychiatric disorders) | 0 (0) | 1 (1) — Worsening Depression
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Atomoxetine (N=18) | Matching Placebo (N=20)
Weight Loss (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Appetite Loss (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Xerostomia (Gastrointestinal disorders) | 7 (7) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2)
Insomnia (Nervous system disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Difficulty Urinating (Renal and urinary disorders) | 2 (2) | 0/0 (0)
Urine Retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
We cannot rule out carryover effects. Additionally, the sample size may be too low to detect small treatment changes, the treatment duration may have been too brief, and our participants had only early-stage HD which may have limited the drug effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes